CLINICAL TRIAL: NCT01991626
Title: Evaluation of the Effects of an Exogenous Phytase on Iron Absorption From Lipid Nutrient Supplements Added to Complementary Foods
Brief Title: Evaluation of the Effects of an Exogenous Phytase on Iron Absorption From LNS Added to Complementary Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Fe-LNS
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — 6-Phytase; Iron-Dextran Complex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (10):
- LNS (Other): Maize meal mixed with Lipid Nutrient Supplement (LNS) containing micronutrient powder
  Interventions: Dietary Supplement: micronutrient powder
- FePP-Emulsion mixed (Other): Fat emulsion mixed to the meal containing FePP
  Interventions: Dietary Supplement: Iron pyrophosphate (FePP)
- FeSO4-Mixed (Other): meals containing FeSO4 mixed with a fat emulsion
  Interventions: Dietary Supplement: Iron sulphate
- FePP-Emulsion before (Other): Fat emulsion taken before a meal containing FePP
  Interventions: Dietary Supplement: Iron pyrophosphate (FePP)
- FeSO4- Emulsion before (Other): Fat emulsion taken before a maize meal containing FeSO4
  Interventions: Dietary Supplement: Iron sulphate
- LNS-Phytase (Other): Maize meal mixed with LNS containing micronutrient powder and phytase
  Interventions: Dietary Supplement: micronutrient powder (containing FeSO4), phytase
- phytase (Other): Maize meal containing micronutrient powder and phytase
  Interventions: Dietary Supplement: micronutrient powder (containing FeSO4), phytase
- MNP-control (Other): maize meal containing micronutrient powder (MNP)
  Interventions: Dietary Supplement: micronutrient powder
- FePP control (Other): Maize meal containing FePP
  Interventions: Dietary Supplement: Iron pyrophosphate (FePP)
- FeSO4 control (Other): Maize meal containing FeSO4
  Interventions: Dietary Supplement: Iron sulphate

INTERVENTIONS:
Dietary Supplement: micronutrient powder
  Arms: LNS; MNP-control
Dietary Supplement: micronutrient powder (containing FeSO4), phytase
  Arms: LNS-Phytase; phytase
Dietary Supplement: Iron pyrophosphate (FePP)
  Arms: FePP control; FePP-Emulsion before; FePP-Emulsion mixed
Dietary Supplement: Iron sulphate
  Arms: FeSO4 control; FeSO4- Emulsion before; FeSO4-Mixed

SUMMARY:
Previous studies on iron absorption have focused on the effects on the addition of iron absorption enhancers like ascorbic acid and EDTA to a meal and more recently the enzymatic phytic acid removal through phytase. The investigators want here to investigate the effects of fat on iron absorption with and without the addition of exogenous phytase as a potential iron absorption enhancer in lipid nutrient supplements (LNS) products compared to micronutrient powder(MNP) products.

Furthermore the investigators will evaluate the effects of Lipids- on iron absorption to induce the ileal brake by ingestion of a fat emulsion prior to a meal. Increasing the caloric density of a meal by increasing its fat content might enhance iron absorption by delaying gastric emptying, gastric acid secretion and increasing Fe stomach residence time.

ELIGIBILITY:
Inclusion Criteria:

Reproductive age females 18-45 years

* Normal body mass index (17.5-25 kg/m2)
* No intake of mineral/vitamin supplements 2 weeks before and during the study
* No metabolic or gastrointestinal disorders
* No food allergies or other chronic disorders or eating disorders assessed by self-report
* Having received full oral and written information about the aims and procedures of the study
* Willing to comply with the study procedure
* Having provided oral and written informed consent

Exclusion Criteria:

* Regular intake of medication (except oral contraceptives)
* Blood donation or significant blood loss (accident, surgery) over the past 4 months
* Currently participating in another clinical trial or having participated in another clinical trial during the last 30 days prior to the beginning of this study
* Former participation in a study involving administration of iron stable isotopes
* Subject who cannot be expected to comply with study protocol
* Pregnancy or lactation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Iron bio-availability from Oral Iron Supplements | 14 days
  Iron bioavailability will be assessed with stable isotopic labels. The shift in the isotopic ratio in human whole blood 14 days after administration will be measured with mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Prof, Principal Investigator — ETH Zürich

REFERENCES:
- [Derived] Monnard A, Moretti D, Zeder C, Steingotter A, Zimmermann MB. The effect of lipids, a lipid-rich ready-to-use therapeutic food, or a phytase on iron absorption from maize-based meals fortified with micronutrient powders. Am J Clin Nutr. 2017 Jun;105(6):1521-1527. doi: 10.3945/ajcn.116.142976. Epub 2017 May 3. PMID 28468891